CLINICAL TRIAL: NCT02624414
Title: A Prospective Study of the Feasibility of Capsule Colonoscopy in Crohn's Disease and Its Correlation With Conventional Colonoscopy and Faecal Calprotectin
Brief Title: Capsule Colonoscopy in Crohn's Disease and Its Correlation With Conventional Colonoscopy and Faecal Calprotectin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014.214
Record Dates: First submitted 2015-11-25; First posted 2015-12-08 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti TNF induction therapy 6-12 months (Other): All subjects will be identified through The Royal Melbourne Hospital's IBD clinic, associated specialty clinics and the colonoscopy waiting list of The Royal Melbourne Hospital. The potential participants who have been commenced on Anti TNF induction therapy 6-12 months prior to commencement of the study will be identified. The potential participants identified in this way will be informed of the project at the time of contact and assessment; in some instances the potential participant will be informed of the project via telephone where subjects are remote. The potential participants will be provided an Ethically-approved information sheet at this time. Consent will be gained at the time of assessment.
  Interventions: Device: PillCam® COLON 2 Capsule Endoscopy

INTERVENTIONS:
Device: PillCam® COLON 2 Capsule Endoscopy

SUMMARY:
Aims:

* To study the feasibility of capsule colonoscopy in patients with Crohn's Disease (CD).
* To compare the results of capsule colonoscopy with conventional colonoscopy in assessing mucosal healing.
* To correlate the level of faecal calprotectin with the results of capsule colonoscopy and conventional colonoscopy.
* To document changes in clinical practice attributable to the capsule colonoscopy findings a) concordant with and b) in addition to the parallel findings at colonoscopy and ileoscopy.

Project design: Cross sectional, prospective, comparative study

Methodology: Patients of the Royal Melbourne Hospital (RMH) and other associated speciality clinics with an established diagnosis of CD who need assessment of mucosal healing and have consented to be part of the study will undergo capsule colonoscopy and conventional colonoscopy on the same day after undergoing bowel preparation. The images of both the conventional and capsule colonoscopies will be recorded. In addition calprotectin (an inflammatory marker in faeces) will be measured in a sample of faeces collected by the patients prior to the colonoscopy day.

Professor Macrae and the scholarly selective student researcher will assess the recorded images obtained from capsule colonoscopies once the images have been deidentified.

To assess the level of mucosal disease they will use the Simple Endoscopic Score for CD (SESCD).

The results of the assessment of mucosal healing obtained from conventional colonoscopy will be compared with those of capsule colonoscopy and levels of faecal calprotectin will then be correlated.

ELIGIBILITY:
Inclusion Criteria:

* Adults with established diagnosis of CD with ileal, colonic or ileo-colonic disease aged 18-75 years. Gender: both male and female
* Patients of RMH IBD clinic and other specialty clinics where assessment of mucosal healing is clinically indicated this includes: Patients who have had Anti TNF induction therapy 6-12 months prior to commencement of this study AND/OR Patients referred for colonoscopy to assess mucosal disease status with a view to treatment escalation based on the findings.

Exclusion Criteria:

Patients must not:

* Have known/suspected gastrointestinal obstruction
* Have swallowing disorder
* Have a known oesophageal stricture
* Have severe gastroparesis
* Have dementia
* Have a cardiac pacemaker or other implanted medical device
* Have sever cardiac or renal insufficiency
* Have a previous allergy or contraindication to bowel preparation
* Be pregnant
* Prior major abdominal surgery
* Colonoscopy is contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Assess bowel cleanness based on the % of mucosal surface visualized by the Capsule colonoscopy | 24 months
  The quality of bowel preparation will be assessed using a new grading system proposed by Segal, et al, University of Melbourne Honours thesis in preparation, 2014. The investigator will assess five colonic segments (cecum, ascending, transverse and descending colon and the rectum). The investigator will assess bowel cleanness based on the % of mucosal surface visualized by the capsule for the presence of: Faecal residue, Turbid Fluid, Bubbles , Faecal residue on Dome, Rapid movement , Poor lighting, Light reflection.
  Each segment will be given a number out of 4: 0 =not present and 4=significantly prevented mucosal visualization.
  SES-CD= sum of the above 4 variables for 5 bowel segments (rectum, sigmoid and ascending colon, transverse colon, descending colon and ileum.
  The images taken during this procedure will be recorded and analysed at a later date.
Simple Endoscopic Score for Crohn's Disease from Conventional colonoscopy | 24 months
Levels of Faecal calprotectin | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Finlay Macrae, Principal Investigator — Melbourne Health
Locations (1):
- Royal Melbourne Hospital, Parkville, Victoria, Australia